CLINICAL TRIAL: NCT01430637
Title: Comprehensive Genome Sequencing of Desmoplastic Small Round Cell Tumors
Brief Title: Studying Genes in Samples From Younger Patients With Desmoplastic Small Round Cell Tumor Registered on COG-D9902 or COG-ABTR01B1
Status: Completed | Type: Observational
Sponsor: Children's Oncology Group (Network)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Other Study IDs: ARST11B5; COG-ARST11B5 (Other: Children's Oncology Group); ARST11B5 (Other: Children's Oncology Group); NCI-2011-03455 (Registry Identifier: CTRP (Clinical Trial Reporting Program))
Record Dates: First submitted 2011-09-07; First posted 2011-09-08 (Estimated); Last update posted 2016-05-18 (Estimated); Status verified 2016-05

CONDITIONS: Sarcoma
Keywords: childhood desmoplastic small round cell tumor; metastatic childhood soft tissue sarcoma; nonmetastatic childhood soft tissue sarcoma; recurrent childhood soft tissue sarcoma; recurrent adult soft tissue sarcoma; stage I adult soft tissue sarcoma; stage II adult soft tissue sarcoma; stage III adult soft tissue sarcoma; stage IV adult soft tissue sarcoma; adult desmoplastic small round cell tumor
MeSH Terms: conditions — Sarcoma; Desmoplastic Small Round Cell Tumor | interventions — Gene Expression Profiling; Base Sequence; Polymerase Chain Reaction; Pharmacogenomic Testing

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Genetic: DNA analysis
Genetic: RNA analysis
Genetic: gene expression analysis
Genetic: mutation analysis
Genetic: nucleic acid sequencing
Genetic: polymerase chain reaction
Other: laboratory biomarker analysis
Other: pharmacogenomic studies

SUMMARY:
RATIONALE: Studying samples of blood and tumor tissue from patients with cancer in the laboratory may help doctors learn more about changes that occur in DNA and identify biomarkers related to cancer.

PURPOSE: This research study is studying genes in samples from younger patients with desmoplastic small round cell tumor registered on COG-D9902 or COG-ABTR01B1.

DETAILED DESCRIPTION:
OBJECTIVES:

* To perform whole-exome sequencing on desmoplastic small round cell tumor (DSRCT) samples and their available matched normal samples to identify novel mutations, single nucleotide polymorphisms, or copy number changes associated with these tumors.
* To identify regions of interest that may be involved in the pathogenesis (including the region of EWSR1-WT1 translocation) from the whole-exome sequencing and perform detailed resequencing and transcriptone sequencing to further define the molecular aberrations at the RNA level.

OUTLINE: This is a multicenter study.

Archived tumor tissue samples are analyzed for DNA sequencing, effects of RNA on gene expression levels, novel RNA isoforms, splice variants, and translocations.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Tumor and blood samples from patients registered on COG-D9902 or COG-ABTR01B1 obtained from the Cooperative Human Tissue Network (CHTN) and the Children's Oncology Group (COG) tumor banks
* Matched normal samples

PATIENT CHARACTERISTICS:

* Not specified

PRIOR CONCURRENT THERAPY:

* Not specified

Max Age: 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Study Population: Patients registered on COG-D9902 or COG-ABTR01B1.
Sampling Method: Non-Probability Sample
Enrollment: 20 (Estimated)
Dates: Start 2011-09; Primary Completion 2016-05 (Actual)

PRIMARY OUTCOMES:
Identification of novel mutations, single nucleotide polymorphisms, and copy number changes associated with DSRCT
Identification of genomic regions involved in pathogenesis of DSRCT

CONTACTS AND LOCATIONS:
Overall Officials: Pooja Hingorani, MD, Principal Investigator — Phoenix Children's Hospital